CLINICAL TRIAL: NCT03068468
Title: A Randomized, Double-Blind, Placebo-Controlled, Parallel-Group Study to Evaluate the Efficacy and Safety of Intravenously Administered BIIB092 in Participants With Progressive Supranuclear Palsy
Brief Title: Study of BIIB092 in Participants With Progressive Supranuclear Palsy
Acronym: PASSPORT
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: 251PP301(PASSPORT) primary endpoint was not met;Biogen decision to close the study early. There were no safety concerns with the PASSPORT study.
Sponsor: Biogen (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 251PP301; 2016-002554-21 (EudraCT Number); CN002-012 (Other: Briston-Myers Squibb)
Record Dates: First submitted 2017-02-27; First posted 2017-03-01 (Actual); Results first posted 2020-12-21 (Actual); Last update posted 2020-12-21 (Actual); Status verified 2020-11

CONDITIONS: Supranuclear Palsy, Progressive
MeSH Terms: conditions — Supranuclear Palsy, Progressive | interventions — gosuranemab

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- BIIB092 (Experimental): Participants will receive BIIB092 50 mg/ml intravenous (IV) infusion once every 4 weeks for 48 weeks in double blind treatment period followed by BIIB092 50 mg/ml IV infusion once every 4 weeks starting at Week 52 up to Week 208.
  Interventions: Drug: BIIB092
- Placebo (Placebo Comparator): Participants will receive BIIB092 matching placebo IV infusion once every 4 weeks for 48 weeks in double blind treatment period followed by BIIB092 50 mg/ml IV infusion once every 4 weeks starting at Week 52 up to Week 208.
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: BIIB092 — BIIB092 intravenous infusion on specified days
  Other Names: BMS-986168
  Arms: BIIB092
Drug: Placebo — Placebo intravenous infusion on specified days
  Arms: Placebo

SUMMARY:
The Primary objective of the study is to evaluate the efficacy of BIIB092, compared to placebo, as measured by a change from baseline in the PSP Rating Scale (PSPRS) at Week 52 and to assess the safety and tolerability of BIIB092, relative to placebo, by measuring the frequency of deaths, SAEs, AEs leading to discontinuation, and Grade 3 & 4 laboratory abnormalities.

The Secondary objective of the study is to evaluate the efficacy of BIIB092, compared to placebo, as measured by a change in baseline in the Movement Disorder Society (MDS)-sponsored revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II at Week 52, to evaluate the efficacy of BIIB092, compared to placebo, as measured by the Clinical Global Impression of Change (CGI-C) at Week 52, to evaluate the efficacy of BIIB092, compared to placebo, as measured by a change in baseline in the Repeatable Battery for the Assessment of Neuropsychological Disease Severity (RBANS) at Week 52 and to assess the impact of BIIB092 on quality of life, relative to placebo, as measured by change from baseline on the Progressive Supranuclear Palsy Quality of Life scale (PSP-QoL) at Week 52.

DETAILED DESCRIPTION:
This study, previously posted by Bristol-Myers Squibb, has transitioned to Biogen under a licensing agreement.

ELIGIBILITY:
Key Inclusion Criteria:

* Participants with probable or possible PSP
* Able to ambulate independently or with assistance
* Able to tolerate MRI
* Have reliable caregiver to accompany participant to all study visits
* Score greater or equal to 20 on the Mini Mental State Exam (MMSE) at screening
* Participant must reside outside a skilled nursing facility or dementia care facility at the time of screening and admission to such a facility must not be planned

Key Exclusion Criteria:

* Presence of other significant neurological or psychiatric disorders
* Diagnosis of amyotrophic lateral sclerosis (ALS) or other motor neuron disease
* History of early, prominent rapid eye movement (REM) sleep behavior disorder
* History of or screening brain MRI scan indicative of significant abnormality
* Known history of serum or plasma progranulin level less than one standard deviation below the normal patient mean for the laboratory performing the assay

NOTE: Other protocol defined Inclusion/Exclusion criteria may apply

Ages: 41 Years to 86 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 490 (Actual)
Dates: Start 2017-06-01 (Actual); Primary Completion 2019-09-06 (Actual); Study Completion 2020-02-07 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Biogen
Locations (82):
- United States (29):
  - Research Site, Phoenix, Arizona
  - Research Site, Scottsdale, Arizona
  - Research Site, Sun City, Arizona
  - Research Site, Fountain Valley, California
  - Research Site, La Jolla, California
  - Research Site, Los Angeles, California
  - Research Site, San Francisco, California
  - Research Site, Boca Raton, Florida
  - Research Site, Gainesville, Florida
  - Research Site, Tampa, Florida
  - Research Site, Chicago, Illinois
  - Research Name, Chicago, Illinois
  - Research Site, Indianapolis, Indiana
  - Research Site, Kansas City, Kansas
  - Research Site, New Orleans, Louisiana
  - Research Site, Baltimore, Maryland
  - Research Site, Boston, Massachusetts
  - Research Site, Burlington, Massachusetts
  - Research Site, Farmington Hills, Michigan
  - Research Site, Minneapolis, Minnesota
  - Research Site, New Brunswick, New Jersey
  - Research Site, Albany, New York
  - Research Site, New York, New York
  - Research Site, Hershey, Pennsylvania
  - Research Site, Philadelphia, Pennsylvania
  - Research Site, Charleston, South Carolina
  - Research Site, Dallas, Texas
  - Research Site, Charlottesville, Virginia
  - Research Site, Seattle, Washington
- Research Site, North Melbourne, Victoria, Australia
- Austria (2):
  - Research Site, Innsbruck, Tyrol
  - Research Site, Vienna
- Canada (3):
  - Research Site, London, Ontario
  - Research Site, Ottawa, Ontario
  - Research Site, Toronto, Ontario
- France (7):
  - Research Site, Bordeaux
  - Research Site, Lille
  - Research Site, Marseille
  - Research Site, Nîmes
  - Research Site, Paris
  - Research Site, Rennes
  - Research Site, Toulouse
- Germany (13):
  - Research Site, Munich, Bavaria
  - Research Site, Marburg, Hesse
  - Research Site, Rostock, Mecklenburg-Western-Pommerania
  - Research Site, Düsseldorf, North Rhine-Westphalia
  - Research Site, Dresden, Saxony
  - Research Site, Kiel, Schleswig-Holstein
  - Research Site, Lübeck, Schleswig-Holstein
  - Research Site, Beelitz-Heilstätten
  - Research Site, Bochum
  - Research Site, Bonn
  - Research Site, Essen
  - Research Site, Kassel
  - Research Site, Ulm
- Research Site, Athens, Marousi, Greece
- Italy (3):
  - Research Site, Salerno, Campania
  - Research Site, Pisa
  - Research Site, Venice-Lido
- Japan (7):
  - Research Site, Nagoya, Aichi-ken
  - Research Site, Kamagaya, Chiba
  - Research Site, Sapporo, Hokkaido
  - Research Site, Sagamihara, Kanagawa
  - Research Site, Kodaira, Tokyo
  - Research Site, Yonago, Tottori
  - Research Site, Shizuoka
- Russia (2):
  - Research Site, Krasnoyarsk
  - Research Site, Moscow
- Research Site, Seoul, South Korea
- Spain (6):
  - Research Site, Pamplona, Navarre
  - Research Site, Barakaldo, Vizcaya
  - Research Site, Barcelona
  - Research Site, Madrid
  - Research Site, Seville
  - Research Site, Valencia
- United Kingdom (7):
  - Research Site, Cambridge, Cambridgeshire
  - Research Site, Brighton, East Sussex
  - Research Site, Southampton, Hampshire
  - Research Site, Liverpool, Merseyside
  - Research Site, Newcastle upon Tyne, Tyne and Wear
  - Research Site, Newport, Wales
  - Research Site, London

REFERENCES:
- [Derived] Jaeger J, Yang L, Li Y, Castrillo-Viguera C, Haeberlein SB, Dam T, O'Gorman J. Development of a cognitive composite for measuring change in progressive supranuclear palsy. Parkinsonism Relat Disord. 2021 Nov;92:94-100. doi: 10.1016/j.parkreldis.2021.10.007. Epub 2021 Oct 12. PMID 34736158
- [Derived] Dam T, Boxer AL, Golbe LI, Hoglinger GU, Morris HR, Litvan I, Lang AE, Corvol JC, Aiba I, Grundman M, Yang L, Tidemann-Miller B, Kupferman J, Harper K, Kamisoglu K, Wald MJ, Graham DL, Gedney L, O'Gorman J, Haeberlein SB; PASSPORT Study Group. Safety and efficacy of anti-tau monoclonal antibody gosuranemab in progressive supranuclear palsy: a phase 2, randomized, placebo-controlled trial. Nat Med. 2021 Aug;27(8):1451-1457. doi: 10.1038/s41591-021-01455-x. Epub 2021 Aug 12. PMID 34385707

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Participants were enrolled at 89 investigative sites in the United States, Australia, Austria, Canada, France, Germany, Greece, Italy, Japan, Republic of Korea, Russia Federation, Spain and United Kingdom from June 01, 2017 to February 07, 2020.
Pre-assignment Details: A total of 490 participants with Progressive Supranuclear Palsy disease were enrolled and randomised in the study. Of these, 486 participants received the study drug in placebo-controlled (PC) period. After completing PC period, 416 participants entered and dosed in open-label extension (OLE) period and no participants completed the study due to early termination of the study.
Groups:
- Placebo (PC Period): Participants assigned to BIIB092 matching placebo intravenous (IV) infusion once every 4 weeks for 48 weeks in double blind PC period and receive only placebo.
- BIIB092 2000 mg (PC Period): Participants who received at least one dose of BIIB092 2000 mg and were either assigned to BIIB092 2000 milligrams (mg) IV infusion or BIIB092 matching placebo IV infusion once every 4 weeks for 48 weeks in double blind PC period.
- BIIB092 Late Start (OLE Period): Late start subjects received only placebo in the placebo-controlled period and assigned to BIIB092 2000 mg IV infusion once every 4 weeks starting at Week 52 in the OLE period.
- BIIB092 Early Start (OLE Period): Early start subjects are those who received BIIB092 2000 mg in the placebo-controlled period and assigned to BIIB092 2000 mg IV infusion once every 4 weeks starting at Week 52 in the OLE period.
Period: Placebo-Controlled Period
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period) | BIIB092 Late Start (OLE Period) | BIIB092 Early Start (OLE Period)
Started | 166 | 324 | 0 | 0
Treated | 165 | 321 | 0 | 0
Completed (Participants who completed the study PC period) | 144 | 279 | 0 | 0
Not Completed | 22 | 45 | 0 | 0
Not completed — Randomized but not Treated | 1 | 3 | 0 | 0
Not completed — Lack of Efficacy | 0 | 1 | 0 | 0
Not completed — Adverse Event | 16 | 21 | 0 | 0
Not completed — Withdrawal by Subject | 3 | 11 | 0 | 0
Not completed — Withdrawal by Parent/Guardian | 1 | 2 | 0 | 0
Not completed — Reason Not Specified | 1 | 6 | 0 | 0
Not completed — Death | 0 | 1 | 0 | 0
Period: Open-Label Extension Period
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period) | BIIB092 Late Start (OLE Period) | BIIB092 Early Start (OLE Period)
Started | 0 | 0 | 140 (4 participants did not enter OLE period.) | 276 (3 participants did not enter OLE period.)
Completed | 0 | 0 | 0 | 0
Not Completed | 0 | 0 | 140 | 276
Not completed — Lack of Efficacy | 0 | 0 | 1 | 2
Not completed — Adverse Event | 0 | 0 | 13 | 17
Not completed — Withdrawal by Subject | 0 | 0 | 7 | 20
Not completed — Death | 0 | 0 | 0 | 1
Not completed — Lost to Follow-up | 0 | 0 | 1 | 0
Not completed — Failure to Meet Randomization Criteria | 0 | 0 | 2 | 0
Not completed — Withdrawal by Sponsor | 0 | 0 | 115 | 228
Not completed — Withdrawal by Parent/Guardian | 0 | 0 | 0 | 4
Not completed — Reason not Specified | 0 | 0 | 1 | 4

BASELINE CHARACTERISTICS:
Population: Intent-to-treat (ITT) population included randomized participants who had received at least 1 dose of blinded study treatment (BIIB092 or Placebo).
Groups:
- Total: Total of all reporting groups
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period) | Total
Number analyzed (Participants) | 165 | 321 | 486
Age, Continuous [Mean (Standard Deviation); unit: years] | 68.9 (6.57) | 68.7 (7.02) | 68.7 (6.86)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 74 | 136 | 210
  Male | 91 | 185 | 276
Ethnicity (NIH/OMB) [Count of Participants; unit: Participants]
  Hispanic or Latino | 5 | 7 | 12
  Not Hispanic or Latino | 117 | 242 | 359
  Unknown or Not Reported | 43 | 72 | 115
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Race: White | 138 | 281 | 419
  Race: Black or African American | 1 | 1 | 2
  Race: Asian Indian | 3 | 3 | 6
  Race: Chinese | 0 | 1 | 1
  Race: Japanese | 16 | 23 | 39
  Race: Asian Other | 4 | 10 | 14
  Race: Unknown | 3 | 2 | 5

OUTCOME MEASURES:

1. Primary Outcome: Change From Baseline in Progressive Supranuclear Palsy Rating Scale (PSPRS) at Week 52
Description: The PSPRS is a quantitative measure of disability in participants with PSP. The PSPRS comprises 28 items in 6 areas. Six items are rated on a 3-point scale (0-2) and 22 are rated on a 5-point scale (0-4). The 6 areas are the History/Daily Activities, Mentation, Bulbar, Ocular Motor, Limb Motor, and Gait. The 28-item PSPRS total score ranges from 0 (normal) to 100. Fifteen items are selected to form a 15-item PSPRS and three domains are identified: Gait/Limb function, Ocular Motor, and Bulbar. The total 15-item PSPRS score ranges from 0 (normal) to 52. A positive change from baseline indicates worsening.
Time Frame: Baseline, Week 52
Population: ITT population included randomized participants who had received at least 1 dose of blinded study treatment (BIIB092 or Placebo). 'Number of Participants Analyzed' signifies number of participants who had response on Week 52.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 139 | 278
Score on a scale
  PSPRS: 28 items | 10.6 (0.8) | 10.4 (0.6)
  PSPRS: 15 items | 7.57 (0.52) | 7.29 (0.38)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); 28-item:Adjusted mean for each treatment group, difference with Placebo,95% confidence interval and p-value at each time point were based on a mixed model for repeated measures model (MMRM), with change from baseline in 28-item PSPRS total score as dependent variable and with fixed effects of treatment group, time(categorical), treatment group-by-time interaction, baseline 28-item PSPRS, baseline 28-item PSPRS by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.8483, Mixed model for repeated measures (MMRM); Difference = -0.2, 95% CI 2-sided [-2.0 to 1.6]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); 15-items:Adjusted mean for each treatment group, difference with Placebo,95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in 15-item PSPRS total score as dependent variable and with fixed effects of treatment group, time(categorical), treatment groupby-time interaction, baseline 15-item PSPRS, baseline 15-item PSPRS by time interaction, baseline Color Trails 2 test(<=170 or >170 seconds) and region; Test type: Superiority; p = 0.6503, MMRM; Difference = -0.28, 95% CI 2-sided [-1.50 to 0.94]

2. Primary Outcome: Percentage of Participants With Death, Serious Adverse Events (SAEs), Adverse Events (AEs) and Adverse Events (AEs) Leading to Discontinuation of Drug
Description: AEs: any sign, symptom, or diagnosis/disease that is unfavorable or unintended, that is new, or if pre-existing, worsens in participants administered a pharmaceutical product and that does not necessarily have a causal relationship with this treatment. SAEs: an event that results in death; an event that, in the view of the investigator, places the participant at immediate risk of death (a life-threatening event); an outcome that results in a congenital anomaly/birth defect diagnosed in a child of a participant; an event that requires or prolongs inpatient hospitalization; an event that results in persistent or significant disability/incapacity.
Time Frame: up to 52 weeks
Population: Safety population included all randomized participants who had received at least one dose of study treatment (BIIB092 or Placebo). Participants randomized to Placebo that received at least one dose of BIIB092 2000 mg during the placebo-controlled period will be counted in the BIIB092 2000 mg group for the safety population. Three participants who received BIIB092 in Placebo group were counted in BIIB092 200 mg group.
Measure: Number; unit: Percentage of participants
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 162 | 324
Percentage of participants
  Death | 4.9 | 4.9
  SAEs | 32.1 | 27.2
  AEs | 93.2 | 92.9
  AEs Leading to Discontinuation of Drug | 11.1 | 7.4

3. Secondary Outcome: Change From Baseline in Movement Disorder Society (MDS)-Sponsored Revision of the Unified Parkinson's Disease Rating Scale (MDS-UPDRS) Part II at Week 52
Description: The MDS-UPRDRS Part 2 includes 13 items assessing motor aspects of experiences of daily living (M-EDL) these include speech, saliva and drooling, chewing and swallowing, handwriting, doing hobbies and other activities, eating tasks, tremor, dressing, hygiene, turning in bed, getting out of bed, walking and balance, and freezing. All items have 5 responses with uniform anchors of 0= normal, 1= slight, 2= mild, 3= moderate, and 4= severe. Total score ranges from 0 to 52, higher score indicating severe conditions. A positive change from baseline indicates worsening.
Time Frame: Baseline, Week 52
Population: ITT population included randomized participants who had received at least 1 dose of blinded study treatment (BIIB092 or Placebo). 'Number of Participants Analyzed' signifies total number of participants analyzed in this outcome measure.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 143 | 270
Score on a scale | 6.7 (0.6) | 7.0 (0.4)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MDS-UPDRS as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline MDS-UPDRS, baseline MDS-UPDRS by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.6031, MMRM; Difference = 0.4, 95% CI 2-sided [-1.0 to 1.7]

4. Secondary Outcome: Clinical Global Impression of Change (CGI-C) Scale Score
Description: The CGI-C scale measures the change in the patient's clinical status from a specific point in time. Using a 7-point scale, ranging from 1 (very much improved) to 7 (very much worse), with a score of 4 indicating no change.
Time Frame: Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 138 | 271
Score on a scale | 5.3 (0.1) | 5.2 (0.1)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with CGI-C as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline CGI-S, baseline CGI-S by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.7743, MMRM; Difference = -0.0, 95% CI 2-sided [-0.2 to 0.1]

5. Secondary Outcome: Change From Baseline in Progressive Supranuclear Palsy (PSP)-Cognitive Composite Battery Z-Score at Week 52
Description: The PSP cognitive composite battery is used to identify and characterize abnormal cognitive decline in PSP participants. The PSP cognitive composite battery includes 13 sub-tests in total: 11 tests from the RBANS (only the picture naming is excluded), letter number sequencing test, and phonemic fluency test. Three domains are identified: Memory and learning, Visual-Motor function, and Working memory and Executive. A z-score transformation is applied for each component test at each visit, and the final total composite z-score is the average of the three-domain z-scores. A z-score of 0 is equal to the estimated mean adjusted by age and is considered average for this study population. Lower values are indicative of cognitive decline. A negative change from baseline indicates worsening.
Time Frame: Baseline, Week 52
Population: ITT population included randomized participants who had received at least 1 dose of blinded study treatment (BIIB092 or Placebo). 'Number of Participants Analyzed' signifies the total number of participants analyzed in this outcome measure.
Measure: Mean (Standard Error); unit: z-score
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 134 | 249
z-score | -0.283 (0.032) | -0.245 (0.024)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in PSP-cognitive composite battery as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline PSP-cognitive composite battery, baseline PSP-cognitive composite battery by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.3180, MMRM; Difference = 0.038, 95% CI 2-sided [-0.036 to 0.112]

6. Secondary Outcome: Change From Baseline in Repeatable Battery for the Assessment of Neuropsychological Disease Severity (RBANS) Scale at Week 52
Description: The RBANS provides both a total scale score and scores for 5 different cognitive domains. Specifically, the test measures immediate memory, visuospatial/constructional ability, language, attention, and delayed memory. Scores from all subtests are aggregated into a total composite score. RBANS data were age-normed and analyzed as index scores (also referred to as standard scores), which have a mean of 100 and a standard deviation of 15. Higher scores on each sub measure and index indicate better performance. A negative change from baseline indicates worsening.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 111 | 222
Score on a scale | -3.1 (0.7) | -3.2 (0.5)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in RBANS as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline RBANS , baseline RBANS by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds and region; Test type: Superiority; p = 0.8270, MMRM; Difference = -0.2, 95% CI 2-sided [-1.8 to 1.4]

7. Secondary Outcome: Change From Baseline in Progressive Supranuclear Palsy Quality of Life Scale (PSP-QoL) Score
Description: The PSP-QoL is a patient-reported outcome measure developed specifically for assessing the health-related quality of life in people living with PSP. It is validated 45-item questionnaire and visual analog scale that is comprised of 2 subscales: physical health state (22 items), which covers mobility, dysarthria, dysphagia, visual disturbances, self-care, and activities of daily living, and mental health state (23 items), which covers emotional, cognitive and social functioning. Items are given a 6-reponse option format (No Problem, Slight Problem, Moderate Problem, Marked Problem, Extreme Problem and Not Applicable). The subscale results are derived by summing the respective items for that subscale and transforming the scores into a range of 0 to 100, the higher the scores indicating a greater impact of the disease on the aspect measured. The PSP-QoL also comprises of a Life Satisfaction rating gauge, which is a visual analog scale with a range of 0 (worst) to 100 (best).
Time Frame: Baseline, Week 52
Population: ITT population included randomized participants who had received at least 1 dose of blinded study treatment (BIIB092 or Placebo). 'Number of Participants Analyzed' signifies number of participants who had response on Week 52. 'Number Analyzed' signifies the number of participants who were evaluated for the specified parameter.
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 142 | 264
Score on a scale
  Physical Scale Score | 11.3 (1.5) | 11.2 (1.1)
  Mental Scale Score: number analyzed (Participants) | 140 | 264
  Mental Scale Score | 5.6 (1.4) | 6.1 (1.0)
  Satisfaction With Your Life Today: number analyzed (Participants) | 141 | 264
  Satisfaction With Your Life Today | -3.7 (1.8) | -5.4 (1.3)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Physical scale score: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in PSP-QoL as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for PSP-QoL, baseline PSP-QoL by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.9304, MMRM; Difference = -0.2, 95% CI 2-sided [-3.6 to 3.3]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Mental scale score: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in PSPQoL as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-bytime interaction, baseline for PSP-QoL, baseline PSP-QoL by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.7859, MMRM; Difference = 0.5, 95% CI 2-sided [-2.8 to 3.7]
Statistical Analysis 3: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Satisfaction With Your Life Today: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in PSPQoL as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-bytime interaction, baseline for PSP-QoL, baseline PSP-QoL by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.4297, MMRM; Difference = -1.7, 95% CI 2-sided [-5.8 to 2.5]

8. Secondary Outcome: Change From Baseline in Schwab and England Activities of Daily Living (SEADL) Scale Score at Week 48
Description: The SEADL scale is a means of assessing a person's ability to perform daily activities in terms of speed and independence, with 100% indicating total independence, falling to 0%, which indicates a state of complete dependence. The individual is asked to rate his or her function using an 11-point scale (10% increments), from 100% (completely independent; able to do all chores without slowness, difficulty, or impairment; essentially normal; unaware of any difficulty) to 0% (vegetative functions such as swallowing, bladder and bowels are not functioning; bedridden). A negative change from baseline indicates worsening.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 140 | 277
Score on a scale | -13.7 (1.4) | -11.7 (1.0)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in SEADL as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for SEADL , baseline SEADL by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.2084, MMRM; Difference = 2.0, 95% CI 2-sided [-1.1 to 5.2]

9. Secondary Outcome: Change From Baseline in Clinical Global Impression of Severity (CGI-S) Score at Week 52
Description: The Clinical Global Impression of Severity (CGI-S) Rating evaluates the severity of individual symptoms and treatment response in participants with mental disorders. The CGI-S is a 7-point scale that that requires the clinician to rate the severity of the patient's illness at the time of assessment. A rating of 1 is considered normal, or with the least severe symptoms, a rating of 7 is extremely ill, or the worst symptoms.
Time Frame: Baseline, Week 52
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 140 | 269
Score on a scale | 0.6 (0.1) | 0.6 (0.0)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in CGI-S as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for CGI-S, baseline CGI-S by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.5701, MMRM; Difference = -0.0, 95% CI 2-sided [-0.2 to 0.1]

10. Secondary Outcome: Change From Baseline in Phonemic Fluency Test Score at Week 48
Description: Phonemic fluency is a sensitive test for assessing frontal lobe dysfunction. Participants are given a letter of the alphabet and asked to name as many words as they can that start with that letter in 1 minute. The score for each trial is auto-calculated as follows: Trial 1: Total number of correct responses for the first letter (range 0 to 40); Trial 2: Total number of correct responses for the second letter (range 0 to 40). The total score from the two trials will be used for analysis (range 0 to 80). More number of words correlates to better phonemic fluency. A negative change from baseline indicates worsening.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Deviation); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 141 | 273
Score on a scale | -0.9 (0.4) | 0.0 (0.3)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in Phonemic Fluency Test as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline Phonemic Fluency Test, baseline Phonemic Fluency Test by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.0517, MMRM; Difference = 0.9, 95% CI 2-sided [-0.0 to 1.8]

11. Secondary Outcome: Change From Baseline in Letter-Number Sequencing Test at Week 48
Description: Letter number is a test of working memory which involves ordering a series of up to 8 letters and numbers in which the numbers are repeated back first in order starting with the lowest number, then followed by the letters in alphabetical order. LNS consists of 10 items and each item has 3 trials rated as Incorrect (0) or Correct (1). The LNS total raw score (range 0 to 30) is auto-calculated by summing the 10 individual item scores (range 0 to 3 for each item). Higher number of correct items correlated to better performance and a negative change from baseline indicates worsening.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 139 | 271
Score on a scale | -1.9 (0.4) | -1.1 (0.3)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in Letter Number Sequence as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline Letter Number Sequence, baseline Letter Number Sequence by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.0387, MMRM; Difference = 0.9, 95% CI 2-sided [0.0 to 1.7]

12. Secondary Outcome: Change From Baseline in Color Trails at Week 48
Description: The Color Trails test is a language free version of the Trail Making Test and was developed to allow for broader cross cultural assessment. For Part 1 (color trails test 1), the respondent uses a pencil to rapidly connect circles numbered 1-25 in sequence. For Part 2 (color trails test 2), the respondent rapidly connects number circles in sequence, but alternates between pink and yellow background. The length of time to complete each trial is recorded, along with qualitative features of performance indicative of brain dysfunction, such as near-misses, prompts, number sequence errors, and color sequence errors. Less time indicates better performance. A positive change from baseline indicates worsening.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Seconds
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 143 | 279
Seconds
  Color Trails Test 1 | 16.8 (3.6) | 16.9 (2.7)
  Color Trails Test 2 | 10.6 (2.4) | 10.5 (1.8)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Color Trails Test 1: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in Color trails Test 1 as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for Color Trails Test 1, baseline Color Trails Test 1 by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.9815, MMRM; Difference = 0.1, 95% CI 2-sided [-8.1 to 8.3]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Color Trails Test 2: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in Color Trails Test 2 as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for Color Trails Test 2, baseline Color Trails Test 2 by time interaction, and region; Test type: Superiority; p = 0.9869, MMRM; Difference = -0.0, 95% CI 2-sided [-5.7 to 5.6]

13. Secondary Outcome: Change From Baseline in Montreal Cognitive Assessment (MoCA) Score at Week 48
Description: The MOCA was designed as a rapid screening instrument for mild cognitive dysfunction. It assesses different cognitive domains: attention and concentration, executive function, memory, language, visuoconstructional skills, conceptual thinking, calculations, and orientation. Scores on the MOCA range from 0-30, with higher score being better performance. A negative change from baseline indicates worsening.
Time Frame: Baseline, Week 48
Population: as for outcome 3
Measure: Mean (Standard Error); unit: Score on a scale
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 136 | 264
Score on a scale | -1.0 (0.3) | -0.5 (0.2)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MoCA as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for MoCA, baseline MoCA by time interaction,baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.1763, MMRM; Difference = 0.5, 95% CI 2-sided [-0.2 to 1.2]

14. Secondary Outcome: Number of Participants With Treatment Emergent Antibodies (Anti-BIIB092) Positive Results in Serum
Time Frame: Up to Week 48
Population: ADA population - subset of the safety population with at least one evaluable post-baseline evaluable ADA samples.
Measure: Count of Participants; unit: Participants
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 160 | 323
Participants | 7 | 0

15. Secondary Outcome: Change From Baseline of Brain Volumes as Determined by MRI at Week 52
Description: A 3 dimension (3D) T1-weighted MRI was performed to estimate brain volumes (e.g., ventricles, whole brain, midbrain, pons, superior cerebellar peduncle, third ventricle, and frontal lobes).
Time Frame: Baseline, Week 52
Population: Efficacy MRI population is the subset of the ITT population who had a least one measurable brain volumetric measurement. 'Number of Participants Analyzed' signifies number of participants who had response on Week 52. 'Number Analyzed' signifies the number of participants who were evaluated for the specified parameter.
Measure: Mean (Standard Error); unit: Cubic centimeter (cm^3)
Arm/Group | Placebo (PC Period) | BIIB092 2000 mg (PC Period)
Number analyzed (Participants) | 114 | 238
Cubic centimeter (cm^3)
  Ventricles Volume: Change at Week 52: number analyzed (Participants) | 103 | 222
  Ventricles Volume: Change at Week 52 | 3.823 (0.302) | 3.802 (0.216)
  Whole Brain Volume: Change at Week 52: number analyzed (Participants) | 101 | 210
  Whole Brain Volume: Change at Week 52 | -18.612 (1.296) | -19.126 (0.950)
  Midbrain Volume: Change at Week 52: number analyzed (Participants) | 108 | 224
  Midbrain Volume: Change at Week 52 | -0.116 (0.008) | -0.120 (0.006)
  Pons Volume: Change at Week 52: number analyzed (Participants) | 100 | 223
  Pons Volume: Change at Week 52 | -0.198 (0.017) | -0.198 (0.012)
  Cerebellar Peduncle Volume: Change at Week 52: number analyzed (Participants) | 101 | 216
  Cerebellar Peduncle Volume: Change at Week 52 | -0.005 (0.002) | -0.004 (0.002)
  Third Ventricle Volume: Change at Week 52 | 0.140 (0.014) | 0.146 (0.010)
  Frontal Lobe Volume: Change at Week 52: number analyzed (Participants) | 89 | 178
  Frontal Lobe Volume: Change at Week 52 | 1.184 (0.279) | 1.143 (0.205)
Statistical Analysis 1: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Ventricles Volume: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MRI region as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for MRI region, baseline MRI region by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.9527, MMRM; Difference = -0.021, 95% CI 2-sided [-0.726 to 0.684]
Statistical Analysis 2: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Whole Brain Volume: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MRI region as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for MRI region, baseline MRI region by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.7357, MMRM; Difference = -0.514, 95% CI 2-sided [-3.506 to 2.478]
Statistical Analysis 3: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Midbrain Volume: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MRI region as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for MRI region, baseline MRI region by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.6439, MMRM; Difference = -0.004, 95% CI 2-sided [-0.023 to 0.014]
Statistical Analysis 4: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Pons Volume: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MRI region as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for MRI region, baseline MRI region by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.9864, MMRM; Difference = 0.000, 95% CI 2-sided [-0.039 to 0.040]
Statistical Analysis 5: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Cerebellar Peduncle Volume: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MRI region as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for MRI region, baseline MRI region by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.7529, MMRM; Difference = 0.001, 95% CI 2-sided [-0.004 to 0.006]
Statistical Analysis 6: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Third Ventricle Volume: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MRI region as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for MRI region, baseline MRI region by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.6850, MMRM; Difference = 0.006, 95% CI 2-sided [-0.025 to 0.038]
Statistical Analysis 7: Comparison: Placebo (PC Period) vs BIIB092 2000 mg (PC Period); Frontal Lobe Volume: Adjusted mean for each treatment group, difference with Placebo, 95% confidence interval and p-value at each time point were based on an MMRM model, with change from baseline in MRI region as dependent variable and with fixed effects of treatment group, time (categorical), treatment group-by-time interaction, baseline for MRI region, baseline MRI region by time interaction, baseline Color Trails 2 test (<=170 or >170 seconds) and region; Test type: Superiority; p = 0.9000, MMRM; Difference = -0.041, 95% CI 2-sided [-0.680 to 0.598]

ADVERSE EVENTS:
Time Frame: up to 140 weeks
Description: Safety population: randomized participants who had received at least 1 dose of BIIB092 or Placebo. Participants randomized to Placebo that received at least 1 dose of BIIB092 2000 mg during the PC period will be counted in the BIIB092 2000 mg group for the safety population. Total number of participants exposed are participants who received drug in respective study periods. For participants affected, a participant was counted only once within each system organ class/preferred term/study period.
Groups:
- Placebo (Placebo Controlled Period): Participants assigned to BIIB092 matching placebo IV infusion once every 4 weeks for 48 weeks in double blind PC period and receive only placebo.
- BIIB092 2000 mg (Placebo Controlled Period): Participants who received at least one dose of BIIB092 2000 mg and were either assigned to BIIB092 2000 mg IV infusion or BIIB092 matching placebo IV infusion once every 4 weeks for 48 weeks in double blind PC period.
- BIIB092 Late Start (Open-label Extension Period): Late start participants received only placebo in the placebo-controlled period and assigned to BIIB092 2000 mg IV infusion once every 4 weeks starting at Week 52 in the OLE period.
- BIIB092 Early Start (Open-label Extension Period): Early start participants are those who received BIIB092 2000 mg in the placebo-controlled period and assigned to BIIB092 2000 mg IV infusion once every 4 weeks starting at Week 52 in the OLE period.
Arm/Group | Placebo (Placebo Controlled Period) | BIIB092 2000 mg (Placebo Controlled Period) | BIIB092 Late Start (Open-label Extension Period) | BIIB092 Early Start (Open-label Extension Period)
All-Cause Mortality (participants affected / at risk) | 8/162 | 16/324 | 10/137 | 16/279
Serious Adverse Events (participants affected / at risk) | 52/162 | 88/324 | 40/137 | 63/279
Other Adverse Events (participants affected / at risk) | 127/162 | 235/324 | 69/137 | 130/279
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo Controlled Period) (N=162) | BIIB092 2000 mg (Placebo Controlled Period) (N=324) | BIIB092 Late Start (Open-label Extension Period) (N=137) | BIIB092 Early Start (Open-label Extension Period) (N=279)
Anaemia (Blood and lymphatic system disorders) | 0 | 0 | 0 | 1
Iron deficiency anaemia (Blood and lymphatic system disorders) | 1 | 1 | 1 | 0
Acute myocardial infarction (Cardiac disorders) | 0 | 0 | 2 | 0
Atrial fibrillation (Cardiac disorders) | 0 | 0 | 1 | 0
Atrioventricular block complete (Cardiac disorders) | 0 | 0 | 0 | 1
Atrioventricular block second degree (Cardiac disorders) | 1 | 0 | 0 | 0
Cardiac arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Cardiac failure (Cardiac disorders) | 0 | 0 | 0 | 1
Cardio-respiratory arrest (Cardiac disorders) | 0 | 0 | 1 | 0
Hypertensive heart disease (Cardiac disorders) | 1 | 0 | 0 | 0
Myocardial ischaemia (Cardiac disorders) | 0 | 0 | 1 | 0
Colitis microscopic (Gastrointestinal disorders) | 0 | 0 | 1 | 0
Constipation (Gastrointestinal disorders) | 1 | 1 | 0 | 0
Diarrhoea (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Dysphagia (Gastrointestinal disorders) | 5 | 3 | 1 | 4
Faecaloma (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Femoral hernia (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Gastritis (Gastrointestinal disorders) | 0 | 1 | 0 | 0
Hernial eventration (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Hiatus hernia (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Large intestine polyp (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Melaena (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Umbilical hernia (Gastrointestinal disorders) | 0 | 0 | 0 | 1
Upper gastrointestinal haemorrhage (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Volvulus (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Vomiting (Gastrointestinal disorders) | 1 | 0 | 0 | 0
Cyst (General disorders) | 0 | 1 | 0 | 0
Death (General disorders) | 0 | 2 | 1 | 2
Drowning (General disorders) | 0 | 0 | 1 | 0
Euthanasia (General disorders) | 0 | 0 | 0 | 1
Gait disturbance (General disorders) | 0 | 2 | 0 | 0
Gait inability (General disorders) | 0 | 0 | 0 | 1
General physical health deterioration (General disorders) | 1 | 1 | 0 | 0
Multiple organ dysfunction syndrome (General disorders) | 0 | 0 | 1 | 1
Systemic inflammatory response syndrome (General disorders) | 0 | 1 | 0 | 0
Cholelithiasis (Hepatobiliary disorders) | 0 | 1 | 0 | 0
Abscess neck (Infections and infestations) | 1 | 1 | 0 | 0
Bacteraemia (Infections and infestations) | 0 | 0 | 0 | 2
Bacterial infection (Infections and infestations) | 1 | 0 | 0 | 0
Bronchitis (Infections and infestations) | 0 | 1 | 0 | 2
Clostridium difficile colitis (Infections and infestations) | 0 | 0 | 0 | 1
Cystitis (Infections and infestations) | 0 | 1 | 0 | 0
Diverticulitis (Infections and infestations) | 0 | 1 | 0 | 0
Escherichia urinary tract infection (Infections and infestations) | 0 | 0 | 0 | 1
Gastroenteritis (Infections and infestations) | 1 | 0 | 0 | 0
Infection (Infections and infestations) | 1 | 0 | 0 | 0
Influenza (Infections and infestations) | 1 | 1 | 0 | 1
Parainfluenzae virus infection (Infections and infestations) | 0 | 0 | 0 | 1
Pneumonia (Infections and infestations) | 0 | 10 | 5 | 6
Pneumonia influenzal (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary sepsis (Infections and infestations) | 0 | 1 | 0 | 0
Pulmonary tuberculosis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory syncytial virus bronchitis (Infections and infestations) | 0 | 1 | 0 | 0
Respiratory tract infection (Infections and infestations) | 0 | 2 | 0 | 0
Sepsis (Infections and infestations) | 0 | 2 | 1 | 2
Septic shock (Infections and infestations) | 0 | 0 | 1 | 0
Subcutaneous abscess (Infections and infestations) | 1 | 0 | 0 | 0
Urinary tract infection (Infections and infestations) | 3 | 1 | 2 | 4
Urosepsis (Infections and infestations) | 0 | 0 | 0 | 1
Viral infection (Infections and infestations) | 0 | 1 | 0 | 0
Wound infection staphylococcal (Infections and infestations) | 0 | 1 | 0 | 0
Ankle fracture (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Cervical vertebral fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 2
Clavicle fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Concussion (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Contusion (Injury, poisoning and procedural complications) | 1 | 1 | 0 | 0
Craniocerebral injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Facial bones fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Fall (Injury, poisoning and procedural complications) | 10 | 41 | 8 | 11
Femoral neck fracture (Injury, poisoning and procedural complications) | 1 | 3 | 0 | 0
Femur fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 2
Fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Hip fracture (Injury, poisoning and procedural complications) | 0 | 2 | 1 | 0
Human bite (Injury, poisoning and procedural complications) | 0 | 0 | 1 | 0
Humerus fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Joint dislocation (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Lumbar vertebral fracture (Injury, poisoning and procedural complications) | 1 | 0 | 1 | 1
Musculoskeletal foreign body (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Open globe injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 1
Periprosthetic fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Post procedural haemorrhage (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Radius fracture (Injury, poisoning and procedural complications) | 0 | 3 | 0 | 0
Rib fracture (Injury, poisoning and procedural complications) | 1 | 4 | 2 | 0
Road traffic accident (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Scapula fracture (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Skin laceration (Injury, poisoning and procedural complications) | 1 | 4 | 0 | 1
Spinal compression fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 2
Spinal fracture (Injury, poisoning and procedural complications) | 0 | 1 | 1 | 0
Subdural haematoma (Injury, poisoning and procedural complications) | 1 | 2 | 1 | 0
Tendon injury (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tendon rupture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Thermal burn (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Thoracic vertebral fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Tibia fracture (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic haematoma (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Traumatic intracranial haemorrhage (Injury, poisoning and procedural complications) | 0 | 1 | 0 | 0
Wrist fracture (Injury, poisoning and procedural complications) | 1 | 0 | 0 | 0
Wrong dose (Injury, poisoning and procedural complications) | 0 | 0 | 0 | 1
Blood creatine phosphokinase increased (Investigations) | 0 | 0 | 1 | 0
Haemoglobin decreased (Investigations) | 1 | 0 | 0 | 0
Liver function test increased (Investigations) | 0 | 0 | 0 | 1
Lumbar puncture (Investigations) | 0 | 0 | 0 | 1
Dehydration (Metabolism and nutrition disorders) | 0 | 1 | 1 | 1
Diabetes mellitus inadequate control (Metabolism and nutrition disorders) | 1 | 0 | 0 | 0
Failure to thrive (Metabolism and nutrition disorders) | 0 | 2 | 0 | 0
Arthralgia (Musculoskeletal and connective tissue disorders) | 0 | 2 | 0 | 0
Chondrocalcinosis (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Haematoma muscle (Musculoskeletal and connective tissue disorders) | 0 | 1 | 0 | 0
Muscle rigidity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteitis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Osteoarthritis (Musculoskeletal and connective tissue disorders) | 0 | 0 | 0 | 1
Pain in extremity (Musculoskeletal and connective tissue disorders) | 0 | 0 | 1 | 0
Breast cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Breast neoplasm (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Colorectal cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Lung adenocarcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 0 | 0
Malignant melanoma in situ (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Metastatic gastric cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 0 | 1
Pancreatic carcinoma (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 0 | 1 | 1
Pituitary tumour benign (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0 | 0 | 0
Prostate cancer (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1 | 1 | 0
Akathisia (Nervous system disorders) | 0 | 0 | 0 | 1
Cerebral disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Cerebrovascular accident (Nervous system disorders) | 0 | 1 | 0 | 2
Dyskinesia (Nervous system disorders) | 0 | 1 | 0 | 0
Encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Epilepsy (Nervous system disorders) | 0 | 2 | 0 | 0
Lumbosacral radiculopathy (Nervous system disorders) | 1 | 0 | 0 | 0
Metabolic encephalopathy (Nervous system disorders) | 0 | 0 | 0 | 1
Monoparesis (Nervous system disorders) | 0 | 0 | 0 | 1
Movement disorder (Nervous system disorders) | 1 | 0 | 0 | 0
Neurological decompensation (Nervous system disorders) | 0 | 0 | 1 | 0
Noninfective encephalitis (Nervous system disorders) | 1 | 0 | 0 | 0
Peroneal nerve palsy (Nervous system disorders) | 0 | 0 | 1 | 0
Progressive supranuclear palsy (Nervous system disorders) | 3 | 6 | 5 | 4
Seizure (Nervous system disorders) | 0 | 0 | 0 | 2
Somnolence (Nervous system disorders) | 0 | 0 | 1 | 0
Status epilepticus (Nervous system disorders) | 0 | 0 | 1 | 0
Subarachnoid haemorrhage (Nervous system disorders) | 0 | 1 | 0 | 0
Syncope (Nervous system disorders) | 1 | 2 | 1 | 2
Transient ischaemic attack (Nervous system disorders) | 1 | 0 | 1 | 0
Agitation (Psychiatric disorders) | 1 | 0 | 0 | 1
Anxiety (Psychiatric disorders) | 0 | 0 | 0 | 1
Assisted suicide (Psychiatric disorders) | 0 | 0 | 0 | 1
Confusional state (Psychiatric disorders) | 0 | 0 | 0 | 1
Hallucination (Psychiatric disorders) | 0 | 0 | 1 | 0
Insomnia (Psychiatric disorders) | 0 | 0 | 0 | 1
Mental status changes (Psychiatric disorders) | 0 | 1 | 0 | 1
Suicidal ideation (Psychiatric disorders) | 0 | 2 | 2 | 1
Suicide attempt (Psychiatric disorders) | 0 | 2 | 1 | 0
Acute kidney injury (Renal and urinary disorders) | 0 | 2 | 0 | 1
Calculus urinary (Renal and urinary disorders) | 1 | 0 | 0 | 0
Hydronephrosis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Nephrolithiasis (Renal and urinary disorders) | 0 | 1 | 0 | 0
Renal impairment (Renal and urinary disorders) | 0 | 0 | 0 | 1
Ureterolithiasis (Renal and urinary disorders) | 0 | 0 | 0 | 1
Urge incontinence (Renal and urinary disorders) | 1 | 0 | 0 | 0
Urinary retention (Renal and urinary disorders) | 1 | 1 | 0 | 1
Acquired phimosis (Reproductive system and breast disorders) | 1 | 0 | 0 | 0
Benign prostatic hyperplasia (Reproductive system and breast disorders) | 0 | 1 | 0 | 0
Prostatitis (Reproductive system and breast disorders) | 0 | 1 | 0 | 1
Acute respiratory failure (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 1 | 4
Aspiration (Respiratory, thoracic and mediastinal disorders) | 3 | 0 | 1 | 1
Choking (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 1 | 0
Chronic obstructive pulmonary disease (Respiratory, thoracic and mediastinal disorders) | 2 | 1 | 0 | 0
Dyspnoea (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 0
Pleural effusion (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 1 | 0
Pneumonia aspiration (Respiratory, thoracic and mediastinal disorders) | 8 | 6 | 5 | 12
Pneumothorax (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Pulmonary embolism (Respiratory, thoracic and mediastinal disorders) | 0 | 2 | 0 | 1
Pulmonary oedema (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory arrest (Respiratory, thoracic and mediastinal disorders) | 0 | 1 | 0 | 0
Respiratory depression (Respiratory, thoracic and mediastinal disorders) | 0 | 0 | 0 | 1
Respiratory distress (Respiratory, thoracic and mediastinal disorders) | 1 | 0 | 0 | 0
Respiratory failure (Respiratory, thoracic and mediastinal disorders) | 3 | 1 | 0 | 0
Dermal cyst (Skin and subcutaneous tissue disorders) | 1 | 0 | 0 | 0
Aortic aneurysm (Vascular disorders) | 0 | 1 | 0 | 0
Deep vein thrombosis (Vascular disorders) | 0 | 2 | 0 | 1
Haematoma (Vascular disorders) | 1 | 0 | 0 | 1
Orthostatic hypotension (Vascular disorders) | 0 | 1 | 0 | 0
OTHER ADVERSE EVENTS (reported when occurring in more than 5% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Placebo (Placebo Controlled Period) (N=162) | BIIB092 2000 mg (Placebo Controlled Period) (N=324) | BIIB092 Late Start (Open-label Extension Period) (N=137) | BIIB092 Early Start (Open-label Extension Period) (N=279)
Constipation (Gastrointestinal disorders) | 15 | 36 | 4 | 16
Diarrhoea (Gastrointestinal disorders) | 9 | 23 | 4 | 9
Nasopharyngitis (Infections and infestations) | 14 | 28 | 6 | 16
Urinary tract infection (Infections and infestations) | 31 | 56 | 15 | 36
Contusion (Injury, poisoning and procedural complications) | 24 | 41 | 15 | 24
Fall (Injury, poisoning and procedural complications) | 83 | 174 | 45 | 79
Head injury (Injury, poisoning and procedural complications) | 8 | 21 | 4 | 8
Skin abrasion (Injury, poisoning and procedural complications) | 10 | 28 | 7 | 12
Skin laceration (Injury, poisoning and procedural complications) | 18 | 40 | 8 | 14
Arthralgia (Musculoskeletal and connective tissue disorders) | 7 | 18 | 0 | 3
Back pain (Musculoskeletal and connective tissue disorders) | 9 | 15 | 3 | 11
Musculoskeletal pain (Musculoskeletal and connective tissue disorders) | 6 | 19 | 2 | 3
Pain in extremity (Musculoskeletal and connective tissue disorders) | 7 | 17 | 0 | 5
Dizziness (Nervous system disorders) | 13 | 18 | 0 | 3
Headache (Nervous system disorders) | 22 | 31 | 3 | 13
Insomnia (Psychiatric disorders) | 14 | 16 | 4 | 10
Haematoma (Vascular disorders) | 11 | 24 | 7 | 11

LIMITATIONS AND CAVEATS:
Study got terminated as the primary endpoint was not met. PC period was completed at the time of termination. The study was not terminated due to a safety concern.

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
Our agreement is subject to confidentiality but generally the PI can publish, for noncommercial purposes only, results and methods of the trial, but no other Sponsor Confidential Information. PI must give Sponsor no less than 60 days to review any manuscript for a proposed publication and must delay publication for up to an additional 90 days thereafter if Sponsor needs to file any patent application to protect any of Sponsor's intellectual property contained in the proposed publication.

DOCUMENTS (2):
  • Study Protocol (2019-02-04): https://cdn.clinicaltrials.gov/large-docs/68/NCT03068468/Prot_000.pdf
  • Statistical Analysis Plan (2019-11-08): https://cdn.clinicaltrials.gov/large-docs/68/NCT03068468/SAP_001.pdf